CLINICAL TRIAL: NCT05773742
Title: Treatment of Fecal Incontinence and Chronic Constipation With Low-volume Irrigation - Qufora IrriSedo MiniGo
Brief Title: Treatment of Fecal Incontinence and Chronic Constipation With Low-volume Irrigation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 222222
Record Dates: First submitted 2023-02-27; First posted 2023-03-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Constipation; Fecal Incontinence
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-volume irrigation (Experimental): The patients will be instructed to irrigate once daily at a fixed time for 6 weeks. The patients will be instructed to use the irrigation 30 min after breakfast, capitalizing on the gastrocolic response; however, should this not fit in with the individual's lifestyle, then an alternative time of the day may be used. Preferably shortly after a large meal. The patients should fill the pump with 180 milliliters (a full pump) and irrigate with a volume of 160 milliliters of water.
  Interventions: Device: Low-volume irrigation

INTERVENTIONS:
Device: Low-volume irrigation — Qufora IrriSedo MiniGo

SUMMARY:
The aim of this study is to investigate the efficacy of low-volume irrigation on bowel function among patients with fecal incontinence and/or chronic constipation (of heterogenous origin).

DETAILED DESCRIPTION:
The aim of this study is to investigate the efficacy of low-volume irrigation on bowel function among patients with FI and/or CC (of heterogenous origin). Further, the aim is to investigate if low volume irrigation can change the negative impact that symptoms of FI and/or CC (of heterogenous origin) have on the patients' daily activities and QoL. Additionally, the aim is to investigate the short-term and long-term discontinuation rates in relation to treatment with low-volume irrigation. Finally, the aim is to investigate the daily time-consumption, the practical challenges and the side effects related to low-volume irrigation. The study period is six weeks and the participants will be instructed to irrigate once daily with Qufora IrriSedo MiniGo.

This study is an interventional study. Patients with FI and/or CC of heterogenous origin, seen in the Nurse-led Clinic for Bowel Dysfunction at the Pelvic Floor Unit, Aarhus University hospital, will be included. Patients will be offered transanal irrigation as a treatment option. Patients presenting with Bristol stool type 6-7 should be offered conservative treatment to optimize the stool consistency. If patients can be regulated to a Bristol stool type 1-5, they can be invited to participate in the study. If necessary, regulation of the stool consistency in patients presenting with Bristol stool type 1-2 is an option, before introducing transanal irrigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FI, CC or co-existing FI and CC of heterogenous origin.
* Positive Rome IV criteria for constipation and/or positive Rome IV criteria for fecal incontinence.
* Patients with Bristol stool type 1-5 as their primary stool consistency.
* 18 years.
* Ability to understand written and spoken Danish (due to questionnaire validity).

Exclusion Criteria:

* Prior use of transanal irrigation or mini enema.
* Patients with chronic diarrhea (Bristol stool type 6-7).
* Patients with neurogenic bowel dysfunction.
* Participation in research conflicting with the current study.
* Diseases treated with rectal or anal surgery (except minor rectal or anal surgery).
* Physical disability that affects the ability to use QuforaÒ IrriSedo MiniGo.
* Major psychiatric diagnoses.
* Patients with constipation with a chronic opioid use or other medications inducing constipation.
* Pregnancy or plans to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
11-point Likert scale | 6 weeks
  The present bowel functions impact on daily activities (0: no, 10: maximum influence)

SECONDARY OUTCOMES:
11-point Likert scale | 3 months, 6 months, 12 months
  The present bowel functions impact on daily activities (0: no, 10: maximum influence)
11-point Likert scale | 6 weeks, 3 months, 6 months, 12 months
  Assessment of the present bowel function (0: no bowel dysfunction, 10: severe bowel dysfunction)
11-point Likert scale | 6 weeks, 3 months, 6 months, 12 months
  The present bowel functions impact on overall QoL (0: no influence, 10: maximum influence)
11-point Likert scale | 6 weeks, 3 months, 6 months, 12 months
  General satisfaction with present bowel function (0: perfect satisfaction, 10: total dissatisfaction)
11-point Likert scale | 6 weeks, 3 months, 6 months, 12 months
  General satisfaction with current treatment (0: perfect satisfaction, 10: total dissatisfaction)
The St. Mark's fecal incontinence score | 6 weeks, 3 months, 6 months, 12 months
  Participants suffering from fecal incontinence
The Fecal Incontinence Quality of Life Scale | 6 weeks, 3 months, 6 months, 12 months
  Participants suffering from fecal incontinence
PAC-SYM score | 6 weeks, 3 months, 6 months, 12 months
  Participants suffering from constipation
The Patients Assessment of Constipation Quality of life | 6 weeks, 3 months, 6 months, 12 months
  Participants suffering from constipation
The 5-level EQ-5D (EQ-5D-5L) index score | 6 weeks, 3 months, 6 months, 12 months
  For all patients
Discontinuation rates | 6 weeks, 3 months, 6 months, 12 months
  Time until discontinuation and reasons for discontinuation.
Correlation for the primary outcome | 6 weeks
  Correlation between score change in primary outcome and the patients' subjective perception of present bowel function rated on a 11-point Likert scale (0: no bowel dysfunction, 10: severe bowel dysfunction) and the patients' evaluation of the efficacy of low-volume irrigation on bowel function rated on a scale from great improvement to great worsening
Correlation for SMIS and PAC-SYM | 6 weeks
  Correlation between the SMIS or PAC-SYM and the patients' subjective perception of present bowel function rated on a 11-point Likert scale (0: no bowel dysfunction, 10: severe bowel dysfunction) and the patients' evaluation of the efficacy of low-volume irrigation on bowel function rated on a scale from great improvement to great worsening
Practicalities and adverse effects | 6 weeks
  Descriptive analyses of volume and duration of irrigation, efficacy of irrigation with regards to evacuation, practical challenges and adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Mekhael, MD, Study Chair — Aarhus University Hospital; Therese Juul, PhD, Study Chair — Aarhus University Hospital; Klaus Krogh, DMSc, Phd, Study Chair — Aarhus University Hospital; Paul Vollebregt, PhD, MD, Study Chair — Queen Mary University of London/Amsterdam University; Louise Schmidt Grau, MD, Study Chair — Aarhus University Hospital
Locations (1):
- Department of Surgery, Aarhus, Denmark